CLINICAL TRIAL: NCT01950611
Title: Phase II Study to Evaluate the Role of Bortezomib in the Management of Relapsed Acute Promyelocytic Leukemia
Brief Title: Proteasome Inhibition in Acute Promyelocytic Leukemia
Acronym: PIAPL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Vikram Mathews, Professor of Clinical Hematology, Christian Medical College, Vellore, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 8225 27/02/13
Record Dates: First submitted 2013-09-22; First posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Relapsed Acute Promyelocytic Leukemia
Keywords: acute promyelocytic leukemia; arsenic trioxide; proteasome inhibition; bortezomib
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib in treatment (Experimental)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Combination of arsenic trioxide with bortezomib in the treatment of relapsed acute promyelocytic leukemia

SUMMARY:
The clinical outcome of relapsed acute promyelocytic leukemia (APL) is poor with current standard of care approaches. Additionally, standard of care warrants an autologous stem cell transplant to be done once molecular remission is achieved. Unfortunately, the majority of our patients cannot afford this procedure. We have previously reported the clinical outcome of relapsed patients who were managed without a stem cell transplants and showed that the event free survival at 5 years is less than 35%. Pre-clinical data reported from our laboratory demonstrates that there is significant synergy between arsenic trioxide (ATO; which is the accepted standard of care agent for relapsed APL) and Bortezomib (a proteasome inhibitor). We have evaluated this combination extensively in-vitro and this data was accepted as an oral presentation at the American Society of Hematology (ASH) meeting in 2011. More recently we have also reported the potential mechanism for this synergy (Poster at ASH 2012). We also have mouse model data which supports these findings. We plan to move this combination of ATO based therapy combined with Bortezomib to a Phase II clinical trial to validate these observations. The anticipated potential is that we will have a combination therapy that is less expensive, cost effective and safe with comparable clinical outcomes to those treated with the more expensive standard of care which includes an autologous stem cell transplant and which the majority of our patients cannot afford.

ELIGIBILITY:
Inclusion Criteria:

i. Diagnosis of relapsed t(15;17)(PML-RARα) positive APL confirmed by reverse transcriptase polymerase chain reaction (RT-PCR).

ii. Normal cardiac function with normal electrocardiogram (QTc less than 500 msec) within 48 hours of study entry.

iii. Patient or guardian willing to give informed consent / assent. Must not have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.

iv. Patients may have received hydroxyurea, 48 hours or less of all trans retnoic acid (ATRA), and 1 dose of an anthracycline and still be eligible for participation in this study.

v. Life expectancy of at least 2 weeks after entry on study. vi. No age limit for entry into study. vii. ECOG performance score 0, 1, or 2. viii. Fertile patients must agree to use an effective barrier method of contraception (e.g., latex condom, diaphragm, or cervical cap) to avoid pregnancy while on therapy and for 3 years following the discontinuation of therapy.

ix. Have a negative serum or urine pregnancy test prior to the first dose of therapeutic drugs (if patient is a female of childbearing potential). If breast feeding they should be willing to stop breast feeding.

Exclusion Criteria:

i. Intracranial bleed at diagnosis. ii. ECOG performance score 3 and above. iii. Severe uncontrolled infection, fulminant sepsis at diagnosis or documented pneumonia.

iv. History of cardiac arrhythmia; symptomatic coronary heart disease; uncontrollable arterial hypertension (diastolic blood pressure > 115 mm Hg); severe psychiatric disease or other concomitant diseases which do not comply with the criteria for the participation in the study.

v. Acute hepatitis (Bilirubin ≥ 5mg% or liver enzymes ≥ 4 times above laboratory normal value) vi. Acute renal failure or serum creatinine ≥ 2 mg% not reversed by hydration. vii. Patients suffering from an additional malignant tumor. No past history of receiving therapy for another malignancy, apart from squamous cell carcinoma or basal cell carcinoma of the skin.

viii. Pregnancy or lactation. ix. Patients with proven intolerance to the study drugs x. Inability, missing willingness or anticipated lack of compliance by the PI to participate in the study. Must not have any other severe concurrent disease and/or uncontrolled medical conditions, which, in the judgment of the investigator, could predispose patients to unacceptable safety risks or compromise compliance with the protocol.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Safety | 5 years
  Non hematological toxicity to be monitored

SECONDARY OUTCOMES:
Efficacy | 5 years
  1. Proportion of patients that achieve molecular remission at the end of induction
  2. Relapse free, event free and overall survival on long term follow up with this protocol.
  3. Long term toxicity profile of this combination therapy
  4. Duration of cytopenia with this combination in induction
  5. Documentation of support care required and total cost of administering this regimen.
  6. Performance status prior to consolidation therapy, each maintenance course and at the end of the regimen.
  7. Molecular remission status on follow up for 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Haematology, Christian Medical College, Vellore, Tamil Nadu, India

REFERENCES:
- [Derived] Kulkarni U, Ganesan S, Alex AA, Palani H, David S, Balasundaram N, Venkatraman A, Thenmozhi M, Jeyaseelan L, Korula A, Devasia A, Abraham A, Janet NB, Balasubramanian P, George B, Mathews V. A phase II study evaluating the role of bortezomib in the management of relapsed acute promyelocytic leukemia treated upfront with arsenic trioxide. Cancer Med. 2020 Apr;9(8):2603-2610. doi: 10.1002/cam4.2883. Epub 2020 Feb 14. PMID 32059085